CLINICAL TRIAL: NCT00779545
Title: Dose Finding and Dose Regimen Study of Mometasone Furoate Nasal Spray in Perennial Allergic Rhinitis
Brief Title: A Study of Mometasone Furoate Nasal Spray in Perennial Allergic Rhinitis (Study P03748)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03748; JPC-03-342-20
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): The placebo group was divided into 3 groups receiving 1, 2 or 4 sprays/nostril. The regimen of each placebo group was BID
  Interventions: Drug: Placebo
- Mometasone furoate nasal spray 100 mcg QD (Experimental)
  Interventions: Drug: Placebo; Drug: Mometasone furoate
- Mometasone furoate nasal spray 200 mcg QD (Experimental)
  Interventions: Drug: Placebo; Drug: Mometasone furoate
- Mometasone furoate nasal spray 400 mcg QD (Experimental)
  Interventions: Drug: Placebo; Drug: Mometasone furoate
- Mometasone furoate nasal spray 100 mcg BID (Experimental)
  Interventions: Drug: Mometasone furoate
- Mometasone furoate nasal spray 200 mcg BID (Experimental)
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: Placebo — One, two, or four sprays of placebo are administered to the left and right nostrils twice a day (in the morning and at night) for 2 weeks.
  Arms: Mometasone furoate nasal spray 100 mcg QD; Mometasone furoate nasal spray 200 mcg QD; Mometasone furoate nasal spray 400 mcg QD; Placebo
Drug: Mometasone furoate — One spray of mometasone furoate 50 mcg is administered to the left and right nostrils in the morning, and one spray of placebo to the left and right nostrils at night for 2 weeks. The daily dose of mometasone furoate is 100 mcg.
  Other Names: Nasonex; SCH 32088
  Arms: Mometasone furoate nasal spray 100 mcg QD
Drug: Mometasone furoate — Two sprays of mometasone furoate 50 mcg are administered to the left and right nostrils in the morning, and two sprays of placebo to the left and right at night for 2 weeks. The daily dose of mometasone furoate is 200 mcg.
  Other Names: Nasonex; SCH 32088
  Arms: Mometasone furoate nasal spray 200 mcg QD
Drug: Mometasone furoate — Four sprays of mometasone furoate 50 mcg are administered to the left and right nostrils in the morning, and four sprays of placebo to the left and right nostrils at night for 2 weeks. The daily dose of mometasone furoate is 400 mcg.
  Other Names: Nasonex; SCH 32088
  Arms: Mometasone furoate nasal spray 400 mcg QD
Drug: Mometasone furoate — One spray of mometasone furoate 50 mcg is administered to the left and right nostrils twice a day (in the morning and at night) for 2 weeks. The daily dose of mometasone furoate is 200 mcg.
  Other Names: Nasonex; SCH 32088
  Arms: Mometasone furoate nasal spray 100 mcg BID
Drug: Mometasone furoate — Two sprays of mometasone furoate 50 mcg are administered to the left and right nostrils twice a day (in the morning and at night) for 2 weeks. The daily dose of mometasone furoate is 400 mcg.
  Other Names: Nasonex; SCH 32088
  Arms: Mometasone furoate nasal spray 200 mcg BID

SUMMARY:
This is a multicenter, randomized, double-blind within the dose level, parallel group comparison of mometasone furoate nasal spray in subjects with perennial allergic rhinitis to examine the minimal effective dose, the recommended dose, and the dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients of mongoloid race residing in Japan who satisfy all of the following criteria:

  * Patients having symptoms of allergic rhinitis of moderate or severe degree, according to the classification of severity in the guidelines for the treatment of nasal allergy (partial revision) as well as a score of at least 4 in the score of 4 nasal symptoms, at the time of obtaining the informed consent during the pretreatment observation period.
  * Patients in whom the skin or specific IgE test is positive and the cytological examination for eosinophils in nasal discharge or nasal challenge test is positive.
  * Out-patients aged 16 years or over at the time of obtaining the informed consent.
  * Male or female.
  * Patients from whom the informed consent can be obtained in writing (or the informed consent can be obtained from the patient's legally acceptable representative, if under 20 years).
  * Patients who can daily complete the nasal allergy diary.

Exclusion Criteria:

* Patients who meet any of the following exclusion criteria are not included in the present study:

  * Patients with a complication of tuberculous disease or lower respiratory tract infection, or patients with a complication of acute upper respiratory tract inflammation or acute laryngopharyngitis which the (sub) investigator considers necessary to treat at the time of enrollment in the treatment.
  * Patients with a complication of infection or systemic mycosis for which no effective antibiotics are available.
  * Patients with unhealed nasal septum ulcer, nasal surgery, or nasal trauma.
  * Patients with hypersensitivity to steroids and mometasone furoate.
  * Patients who are pregnant, nursing, or possibly pregnant, or who desire to become pregnant during the study period.
  * Patients with severe hepatic, renal, or cardiac disorder, blood disease, diabetes, hypertension, or other serious complication, suffering from problems with systemic condition.
  * Patients in whom pollen is an overlapping allergen and the study is planned to be implemented in the pollen release season.
  * Patients with a complication of vasomotor rhinitis or eosinophilic rhinitis.
  * Patients with a complication of nose disease which may interfere with efficacy evaluation of the investigational product.
  * Patients who were complicated by acute upper respiratory tract inflammation during the 7-day observation period prior to enrollment which may affect the nasal symptoms.
  * Patients who have previously received mometasone furoate nasal spray.
  * Patients who have participated in clinical trial of other investigational product(s) within 4 months before obtaining the informed consent or are participating at present.
  * Patients in whom prior medication effective against allergic rhinitis was withdrawn not long enough before initiation of treatment with the investigational product or the preceding medication cannot be withdrawn.
  * Patients who are being treated with specific desensitization therapy or nonspecific allassotherapy or in whom such the therapy was withdrawn within 3 months before obtaining the informed consent (except for patients receiving the maintenance therapy at present in whom the therapy began more than 6 months before obtaining the informed consent).
  * Other patients whom the (sub) investigator judged to be inappropriate for participation in the present study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2004-04-08 (Actual); Primary Completion 2004-08-06 (Actual); Study Completion 2004-08-06 (Actual)

PRIMARY OUTCOMES:
Change in 4 nasal symptom score (sneezing attack, rhinorrhea, nasal congestion, and nasal itching) from baseline at Week 2 | After 2 weeks of treatment

SECONDARY OUTCOMES:
Change in each nasal symptom (sneezing attack, rhinorrhea, nasal congestion, and nasal itching) | After 1 and 2 weeks of treatment
Overall improvement | After 1 and 2 weeks of treatment
QOL score | At initial day of treatment and after 2 weeks of treatment
Adverse events | From initial day of treatment until 7-10 days after treatment is stopped.
Laboratory tests | From initial day of treatment until treatment is stopped.